CLINICAL TRIAL: NCT03736486
Title: Mil Familias- Santa Barbara Operational Pilot
Brief Title: Mil Familias-Santa Barbara's Operational Pilot to Understand Diabetes in the Latino Community
Acronym: MilFamilias
Status: Completed | Type: Observational
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-5864
Record Dates: First submitted 2018-10-30; First posted 2018-11-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Type2 Diabetes Mellitus; Cardiovascular Diseases
Keywords: Type 2 diabetes; Cardio-metabolic disease; Latino; Hispanic; Especialista
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, Plasma, Buffy coat (white cells)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetes: Male and female adults of Hispanic and/or Latino heritage with an established diagnosis of Type 2 diabetes.

SUMMARY:
The Mil Familias Program is a 10-year initiative to reduce the burden of cardio-metabolic disease among Latino families in the Central Coast of California. The Mil Familias Program involves enrolling 1000 Latino families with at least one member in the family having type 2 diabetes, measuring the 5 determinants of human health: genetics, biology, behavior, psychology and environment, training Latino community health workers ("Especialistas") , creating a Living Information (bio)Bank and planning culturally-relevant interventions.

DETAILED DESCRIPTION:
The Mil Familias Pilot Study aims to develop, operationalize and refine methods to both recruit and collect data from 100 adult participants pertaining to the 5 determinants of human health: genetics, biology, behavior, psychology and environment. Specially-trained Latino and bilingual community health workers known as "Especialistas" will be used to help gather data and to serve as the participants trustworthy health companion. Over 100 variables of information pertaining to the 5 determinants of human health (as listed above) will be gathered and stored to create a Living Information (bio)Bank particular to Latinos. The ultimate goal of this research is to provide the target population with effective, culturally-relevant interventions that are geared toward population specific needs.

ELIGIBILITY:
Inclusion criteria:

1. Males or females ≥ 18 years of age at Visit 1 (screening and enrollment).
2. Self-reported Hispanic and/or Latino heritage.
3. Currently residing in Santa Barbara County, California.
4. Established diagnosis of Type 2 diabetes for at least one year prior to enrollment date.
5. Signed and dated written informed consent by the date of Visit 1.
6. Based on the research staff's judgment, subject must have a good understanding, ability, and willingness to adhere to the protocol, including performance of self-monitored data collection during the wearable device portion.

Exclusion Criteria:

1. Diagnosed severe cardiovascular disease, within the 6 months prior to enrollment Visit 1, defined as: previous stroke; decompensated heart failure New York Heart Association class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty.
2. Life expectancy < 2 years.
3. Any active clinically significant disease or disorder, which in the investigator's opinion could interfere with the participation of the trial.
4. Mental incapacity, psychiatric disorder, unwillingness or language barriers precluding comprehension of study activities and informed consent.
5. Participation in other trials involving medication or device within 1 month prior to Visit 1.
6. Known or suspected abuse of alcohol, narcotics, or illicit drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 125 individuals may be screened and enrolled with the prediction of 20% screen-fail or dropout and 100 people completing SB1K Phase I.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Success (evaluated by Yes/No format) recruiting and establishing a pilot cohort of 100 Latino adults with Type 2 Diabetes and creating data collection methods to describe genetics, biology, behavior, psychology, & environment in Type 2 Diabetes | 1 year
  Mil Familias Program Pilot will measure genetic influences by a family medical history & biobank blood samples. Biologic influences will include laboratory blood draw, physical exam with vital signs & waist circumference measurement, and complete medical & medication history with female menopause, pregnancy, & gestational diabetes status. Behavior influences will include sleep, stress, drug abuse, and diabetes self-assessment management questionnaires. Wearable devices will measure physical activity. Psychological influences will include Patient Health Questionnaire-9, Brief Perceived Ethnic Discrimination Questionnaire Community Version, and Short Form Health Survey. Social/environmental influences will include socio-demographics, Brief Acculturation Scale for Hispanics, personal opinions about type 2 diabetes, and questionnaires [Short Assessment of Health Literacy, Trust in Physician, Health Leads Screening Toolkit, and U.S. Household Food Security Survey].

SECONDARY OUTCOMES:
Socio-demographics measured by questionnaire - including age, gender, race/ethnicity, contact information, number in household, income, education, marital status, occupation, insurance status, immigration status, alcohol & tobacco use, and birth place | Beginning of study - Baseline visit 1
  Socio-demographics assessed by questionnaire.
Self-assessment of diabetes management measured by the American Diabetes Association questionnaire, Participant Self-Assessment of Diabetes Management | Beginning of study - Baseline visit 1
  Participant report and self-assessment of diabetes management by questionnaire
Food security assessed by U.S. Household Food Security Survey Module: Six-item short form | Beginning of study - Baseline visit 1
  Food security or insecurity assessed by a six-item short form developed by the Economic Research Service, United States Department of Agriculture (USDA), September 2012
Social needs screening assessed by the Health Leads Screening Toolkit | Beginning of study - Baseline visit 1
  The Health Leads Screening Tookit (Boston, MA) will be used to determine social needs
Number of visits to a healthcare provider in the last year and difficulty in traveling to a healthcare provider measured by electronic medical record and interview | Beginning of study - Baseline visit 1
  Number of healthcare visits assessed in medical record review and the difficulty in traveling to the healthcare provider assessed by questionnaire
Personal opinion regarding type 2 diabetes burden on Latinos measured by 3 questions - why is diabetes common in Latinos, what can be done to prevent diabetes in Latinos, and what things make it difficult to get help with diabetes when it is needed? | Beginning of study - Baseline visit 1
  Questions regarding personal opinions regarding the burden of diabetes on Latinos measured by specific questions
Support for diabetes care measured by questionnaire adapted from the American Diabetes Association Participant Self-Assessment of Diabetes Management questionnaire | Beginning of study - Baseline visit 1
  How well a participant is supported in diabetes care measured by a questionnaire from the American Diabetes Association (ADA) Participant Self-Assessment of Diabetes Management questionnaire
Medical history, family medical history, and medication status and history assessed by interview and electronic medical records | Day 1 of Visit 2
  Medical history, family medical history, and current medications and medication history assessed by interview and electronic medical records
Menopausal status, pregnancy status, and gestational diabetes history for women determined by interview and electronic medical records | Day 1 of Visit 2
  Menopausal status, pregnancy status, and gestational diabetes history for female participants will be determined by interview and electronic medical records
Measurement by composite physical exam - height, weight, waist circumference, blood pressure, temperature, heart rate & rhythm, and foot examination including questions about neuropathy and retinopathy and dental & eye exams | Day 1 of Visit 2
  Physical exam with vital signs and questions about neuropathy, retinopathy, dental, and eye exams
Composite lab tests: C-Peptide, C-reactive protein, Complete blood count, Comprehensive metabolic panel, Glutamic Acid Decarboxylase (GAD) antibodies, HbA1c, Insulin autoantibody, Lipid panel, Insulin, and Thyroid function | Day 1 of Visit 2
  Laboratory blood draw for evaluation of physiological markers related to diabetes
Microalbumin, creatinine, and microalbumin/creatinine ratio measured in a urine sample | Day 1 of Visit 2
  Urine sample collected for measuring microalbumin, creatinine, and the microalbumin/creatinine ratio
Depression measured by the Patient Health Questionnaire-9 | Day 1 of Visit 2
  The Patient Health Questionnaire (PHQ)-9 is the Major Depressive Disorder (MDD) module of the full PHQ
Drug abuse measured by the Drug Abuse Screening Test (DAST) - 20 | Day 1 of Visit 2
  The purpose of the DAST-20 is to provide a brief, simple, practical, but valid method for identifying individuals who are abusing psychoactive drugs; and to yield a quantitative index score of the degree of problems related to drug use and misuse
Physical activity measured by two wearable physical activity monitors for 1 week | 1 week
  Participants wear an ActiGraph and Fitbit activity monitors simultaneously for 1 week
Acculturation measured by the Brief Acculturation Scale for Hispanics (BASH) | Day 1 of Visit 3
  BASH is a participant reported questionnaire to measure acculturation
Health literacy measured by the Short Assessment of Health Literacy (SAHL) | Day 1 of Visit 3
  SAHL is a participant reported questionnaire to measure health literacy
Perceived Ethnic Discrimination measured by the Brief Perceived Ethnic Discrimination Questionnaire - Community version (PEDQ-CV) | Day 1 of Visit 3
  PEDQ-CV is a participant reported questionnaire to measure perceived ethnic discrimination
Stress measured by the 4 item Perceived Stress Scale (PSS) | Day 1 of Visit 3
  PSS is a participant reported questionnaire to measure stress
Quality of life measured by the Short Form Health Survey (SF-12) | Day 1 of Visit 3
  The SF-12 is a participant reported questionnaire to measure quality of life
Sleep quality measured by the Oviedo Sleep Questionnaire (OSQ) | Day 1 of Visit 3
  The OSQ is a participant reported questionnaire to measure sleep quality
Trust in physician measured by the Trust in Physician (TPS) questionnaire | Day 1 of Visit 3
  The TPS is a questionnaire and scale to determine trust in the physician

OTHER OUTCOMES:
Engagement of a local consortium of partners to implement participant recruitment; data collection, storage, and analysis; healthcare access; and/or intervention measured by the number of major operational partnerships with formal agreements | 1 year
  A local consortium of partners will be engaged with formal operational partnerships that include signed agreements and statements of work. These partnerships will include local health clinics and providers, the county, Hispanic/Latino community groups, other non-profit groups involved with the Hispanic/Latino community, and health promoters such as the Young Men's Christian Association (YMCA).
Success measured by the number of health care workers trained, upskilled, and employed to be community health care workers (Especialistas) and the number of participant encounters with a trained health care worker | 1 year
  Curricula will be developed, delivered, and evaluated by the number of health workers trained & employed and the number of encounters between participants & trained health workers (Especialistas). Three modules of training curriculum will be developed for Type 2 Diabetes (T2D) Educators, Researchers, and Care Navigators. Training includes T2D clinical aspects, health determinants, diabetes education for Latinos, technology integration into diabetes education, focused diabetes education, research fundamentals, Good Clinical Practice, human subjects protections, participant recruitment, selection & enrollment, clinical data collection, qualitative data collection methods, technology to enhance & facilitate diabetes research, health care sequence, diabetes resources, social and health care resources, health insurance coverage & eligibility, making referrals to resources, sociocultural insight to diabetes care navigation, and technology facilitate access to resources.

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, M.D., Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in publications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available after the primary publication of each analysis.
Access Criteria: Data Sharing Agreements will be formulated by a committee of study investigators and community and industry partners.
URL: http://www.milfamilias.com

REFERENCES:
- [Derived] Glantz NM, Morales JM, Bevier WC, Larez A, Hoppe CB, Duncan I, Mackenzie A, Kerr D. Insurance Status and Biological and Psychosocial Determinants of Cardiometabolic Risk Among Mexican-Origin U.S. Hispanic/Latino Adults with Type 2 Diabetes. Health Equity. 2020 May 4;4(1):142-149. doi: 10.1089/heq.2019.0119. eCollection 2020. PMID 32440613
- [Derived] Bevier W, Glantz N, Hoppe C, Morales Glass J, Larez A, Chen K, Kerr D. Self-reported and objectively measured physical activity levels among Hispanic/Latino adults with type 2 diabetes. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e000893. doi: 10.1136/bmjdrc-2019-000893. PMID 32169933